CLINICAL TRIAL: NCT01179204
Title: Is Preoperative Pain Response Upon Tonic Heat Stimulation Predictive for Pain After Total Knee Arthroplasty?
Brief Title: Prediction of Pain in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: H-2-2010-052
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood-samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patiens operated with TKA
  Interventions: Procedure: Preoperative heat stimulation

INTERVENTIONS:
Procedure: Preoperative heat stimulation — Preoperative short and long tonic heat stimulation

SUMMARY:
In this consecutive, prospective cohort study trial the investigators evaluate if preoperative pain response upon heat stimulation is predictive for acute and subacute postoperative pain after total knee arthroplasty.

DETAILED DESCRIPTION:
The preoperative heat stimulation consists of short and long tonic heat stimulation. Pain response is evaluated with an electronic visual analog scale.

Furthermore the investigators evaluate other factors possibly predictable for acute and subacute postoperative pain after total knee arthroplasty - demographic factors, preoperative pain related factors, psychosocial factors (Hospital Anxiety and Depression Scale and Pain Catastrophizing Scale).

ELIGIBILITY:
Inclusion Criteria:

* Ethnic danes, above 18 years and able to give informed consent scheduled for primary, unilateral total knee arthroplasty.

Exclusion Criteria:

* Bilateral / revision arthroplasty
* Disease affection central or peripheral nerve function
* Alcohol and medical abuse
* Daily use of opioids or glucocorticoids
* Malignancy
* BMI > 40
* Depression
* Dementia or other cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated with total knee arthroplasty (TKA)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Cumulated pain (from 0-24 hours after surgery) | 24 hours
  Pain during walk 5 m (VAS)

SECONDARY OUTCOMES:
Cumulated pain (from day 1 to day 7 after surgery) | 7 days
Pain at day 14 after surgery | 14 days
Pain at day 30 after surgery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Troels H. Lunn, M.D, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark